CLINICAL TRIAL: NCT07358507
Title: Investigation of the Effects of Nerve Gliding Exercises on Pain, Function, Joint Position Sense and Weight-Bearing Tolerance in Patients With Ulnar-Sided Wrist Pain
Brief Title: EFFECTS OF NERVE GLIDING EXERCISES ON ULNAR-SIDED WRIST PAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: Ankara University (Other)
Responsible Party: Principal Investigator, Ceren Zorluogullari, Master's Student, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-1761
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Ulnar Wrist Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants in this group will receive standard treatment consisting of patient education, activity modification, massage, and ice application for 4 weeks.
  Interventions: Other: Conventional Physiotherapy
- Mobilization Group (Experimental): Participants in this group will receive standard treatment including patient education, activity modification, massage, and ice application. In addition, they will perform ulnar nerve gliding exercises for 4 weeks.
  Interventions: Other: Ulnar Nerve Gliding Exercises; Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Ulnar Nerve Gliding Exercises — Ulnar nerve gliding exercises will be performed twice a week in the clinic for 4 weeks. Participants will also perform these exercises as a home program 3 times daily.
  Arms: Mobilization Group
Other: Conventional Physiotherapy — Includes patient education, activity modification, classic massage along the ulnar nerve trace, and ice application (10-12 minutes) at the end of each session.

SUMMARY:
The purpose of this study is to learn if adding specific "nerve gliding" exercises to a standard physical therapy program helps reduce pain and improve hand function in people with ulnar-sided (pinky side) wrist pain.

Participants who have had wrist pain for at least 3 months will be randomly assigned to one of two groups. Both groups will receive a standard treatment program that includes patient education, activity modification, massage, and ice application. One group will also perform specific nerve gliding exercises for the ulnar nerve.

Researchers will evaulate pain level, hand function, strength, weight-bearing tolerance, and joint position sense at the beginning and after 4 weeks of treatment to see if the exercises provide extra benefit. The study treatment period lasts for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age.
* History of ulnar-sided wrist pain lasting for at least 3 months.
* Diagnosis of ulnar-sided wrist pain confirmed by a hand surgeon, which may include: fractures or dislocations of the 4th and 5th metacarpals, hamate, triquetrum, lunate, pisiform, distal ulna, or distal radius; Lunotriquetral ligament tears; Kienböck's disease; Ulnar impaction syndrome; Triangular Fibrocartilage Complex (TFCC) injury; carpal instabilities; DRUJ instability; pisotriquetral arthritis; DRUJ arthritis; extensor carpi ulnaris (ECU) tendon subluxation; or tendinitis of the ECU, extensor digiti minimi, and flexor carpi ulnaris.
* Adequate cognitive level (scoring 22 or above on the Montreal Cognitive Assessment scale).

Exclusion Criteria:

* Presence of other diseases involving the hand and wrist (e.g., carpal tunnel syndrome, Dupuytren's disease).
* History of traumatic injury to the hand, wrist, and/or forearm within the last 3 months.
* History of surgery on the hand, wrist, and/or forearm within the last 6 months.
* Currently receiving treatment for hand and wrist problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Pain Level | From enrollment to the end of treatment at 4 weeks
  Pain level will be evaluated using the Visual Analog Scale (VAS) for pain at rest, during activity, and at night.

SECONDARY OUTCOMES:
Wrist Function | Baseline and 4 weeks.
  Patient-Rated Wrist Evaluation (PRWE) questionnaire (0-100 scale, higher scores indicate greater disability)
Grip Strength | Baseline and 4 weeks
  Measured with a Jamar hydraulic hand dynamometer in kg (average of 3 trials)
Wrist Strength | Baseline and 4 weeks
  Wrist flexion and extension strength will be measured with handheld dynamometer.
Weight Bearing Tolerance | Baseline and 4 weeks
  Measured in kg using an analog scale where participants apply maximum force with the wrist.
Joint Position Sense | Baseline and 4 weeks.
  Measured as degrees of deviation from a 30° target position using a goniometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Health Sciences Faculty Physiotherapy and Rehabilitation Department, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No